CLINICAL TRIAL: NCT00920491
Title: BANC4 (BASEL NON - SPECIFIC COMPLAINTS 4) Biomarker-enhanced Disposition Decisions
Brief Title: Biomarker-enhanced ED Disposition Decisions
Acronym: BANC4
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: ED UHBS
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Non-specific Complaints
Keywords: Chief complaint; non-specific symptoms; general weakness / general deterioration; risk assessment in ED patients with non-specific symptoms
MeSH Terms: conditions — Asthenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood (MR-proADM)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with non-specific complaints: patients who do not have specific presenting symptoms (e.g. dyspnea, chest pain etc.)
  Interventions: Biological: biomarker-enhanced disposition decision with proADM

INTERVENTIONS:
Biological: biomarker-enhanced disposition decision with proADM — To compare the outcome of standard of care with an approach combining the standardized course and biomarker levels (biomarker-enhanced disposition decision with proADM) for the disposition of patients with non-specific complaints presenting to the emergency department (ED), in order to evaluate safety.

SUMMARY:
Patients presenting to emergency departments (ED) with non-specific complaints (NSC) such as "not feeling well", "feeling weak", "being tired", "general deterioration" are a very common and well-known, but poorly studied patient group. The differential diagnosis of NSC is extremely broad ranging from insufficient home care to acute life-threatening conditions. Therefore, the evaluation and diagnostic work-up of these mostly elderly patients with NSC is very time-consuming and not straight-forward. Furthermore, the assessment is complicated by comorbidities, polypharmacy or an altered mental status. For this reason, potentially unnecessary diagnostic efforts are undertaken in order to exclude a serious underlying condition, leading to prolonged throughput times and ED observation unit stays.

On the other hand, the patients' condition might be underestimated by ED physicians, which may result in ineffective, delayed or inadequate disposition, as well as poor patient outcomes. BANC (formerly BAUCAS) is a series of clinical studies with the intention to investigate the usefulness of clinical findings and biomarker levels combined for disposition of patients with non-specific complaints presenting to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* All adult non-trauma patients with an Emergency Severity Index (ESI) of 2 or 3 are screened for inclusion

Exclusion Criteria:

* patients with specific chief complaints are excluded. Moreover, patients in whom an unambiguous and clear working hypothesis with logical management steps can be established are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The protocol of the BANC study specifies that patients are consecutively enrolled in order to obtain a random sample of the source population of ED self-referred and referred patients with UC
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
serious condition (potentially life-threatening or requiring early intervention to prevent health status deterioration) | 30 days

SECONDARY OUTCOMES:
30 day mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Nickel CH, Kuster T, Keil C, Messmer AS, Geigy N, Bingisser R. Risk stratification using D-dimers in patients presenting to the emergency department with nonspecific complaints. Eur J Intern Med. 2016 Jun;31:20-4. doi: 10.1016/j.ejim.2016.03.006. Epub 2016 Apr 1. PMID 27053291
- [Derived] Nickel CH, Messmer AS, Ghanim L, Ilsemann-Karakoumis J, Giersdorf S, Hertel S, Ernst S, Geigy N, Bingisser R. Adrenomedullin for Risk Stratification of Emergency Patients With Nonspecific Complaints: An Interventional Multicenter Pilot Study. Medicine (Baltimore). 2016 Jan;95(1):e2395. doi: 10.1097/MD.0000000000002395. PMID 26735540
- [Derived] Karakoumis J, Nickel CH, Kirsch M, Rohacek M, Geigy N, Muller B, Ackermann S, Bingisser R. Emergency Presentations With Nonspecific Complaints-the Burden of Morbidity and the Spectrum of Underlying Disease: Nonspecific Complaints and Underlying Disease. Medicine (Baltimore). 2015 Jul;94(26):e840. doi: 10.1097/MD.0000000000000840. PMID 26131835
- [Derived] Peng A, Rohacek M, Ackermann S, Ilsemann-Karakoumis J, Ghanim L, Messmer AS, Misch F, Nickel CH, Bingisser R. The proportion of correct diagnoses is low in emergency patients with nonspecific complaints presenting to the emergency department. Swiss Med Wkly. 2015 Mar 5;145:w14121. doi: 10.4414/smw.2015.14121. eCollection 2015. PMID 25741894
- [Derived] Nickel CH, Ruedinger JM, Messmer AS, Maile S, Peng A, Bodmer M, Kressig RW, Kraehenbuehl S, Bingisser R. Drug-related emergency department visits by elderly patients presenting with non-specific complaints. Scand J Trauma Resusc Emerg Med. 2013 Mar 5;21:15. doi: 10.1186/1757-7241-21-15. PMID 23497667
- [Derived] Ruedinger JM, Nickel CH, Maile S, Bodmer M, Kressig RW, Bingisser R. Diuretic use, RAAS blockade and morbidity in elderly patients presenting to the Emergency Department with non-specific complaints. Swiss Med Wkly. 2012 May 9;142:w13568. doi: 10.4414/smw.2012.13568. eCollection 2012. PMID 22573483